CLINICAL TRIAL: NCT05329194
Title: A Multicenter, Single-arm, Open-label, Post-Authorization, Phase 4 Effectiveness and Safety Study of Tezepelumab in Adult and Adolescent Participants With Severe Asthma Including Several Under-Studied Populations in the United States (PASSAGE)
Brief Title: Effectiveness and Safety Study of Tezepelumab in Adults & Adolescent Participants With Severe Asthma in the United States
Acronym: PASSAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5180C00032
Record Dates: First submitted 2022-03-17; First posted 2022-04-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Asthma
Keywords: Inhaled corticosteroids (ICS); Post-Authorization; Baseline Blood eosinophil count (BEC); long-acting- β2 Agonist (LABA); Real-world participant population
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tezepelumab (Experimental): Participants will be receiving 210 mg of tezepelumab every 4 weeks (Q4W) from Week 0 until Week 48.
  Interventions: Drug: Tezepelumab

INTERVENTIONS:
Drug: Tezepelumab — Participants will be receiving subcutaneous injection of tezepelumab.
  Other Names: AMG 157 or MEDI9929

SUMMARY:
To asses effectiveness and safety of tezepelumab in adult and adolescent participants with severe asthma including several under-studied populations in the United States.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, open-label, Post-authorization, Phase 4 study to assess the effectiveness of tezepelumab in the United States (US) among a real-world population of adults and adolescent participants with asthma requiring medium-dose to high-dose inhaled corticosteroids (ICS), with additional controller(s) for at least 12 months with documented history of at least 2 asthma exacerbations during the year prior to enrolment. The total duration of the study for each participant will be approximately 56 weeks. Approximately 400 participants will be enrolled. Participants will receive tezepelumab via subcutaneous injection at the study site, over a 48-week treatment period. The study also includes a post-dosing follow-up period from Weeks 48 to 52.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant must be 12 years of age or older, at the time of signing the informed consent form or assent.
* Documented physician-diagnosed asthma for at least 12 months prior to enrollment and confirmed by the Investigator not to be due to alternative diagnoses.
* Documented treatment with medium- to high dose ICS as per Global Initiative for Asthma (GINA) guidelines (GINA 2021) for at least 12 months prior to enrollment.
* Use of additional asthma maintenance controller medication(s) in addition to ICS for at least 12 months prior to enrollment. The additional maintenance controller medication may be contained in a combination product (eg, ICS/ long-acting β-agonist (LABA)).
* Documented history of at least 2 asthma exacerbations during the 12 months prior to enrollment.
* Physician decision that participant is eligible for treatment with tezepelumab according to the approved United States product insert (USPI).
* Currently receiving care from specialist physicians (eg, pulmonologists and/or allergists).
* Provision of signed and dated written informed consent form.

Exclusion Criteria:

* Any contraindication to tezepelumab as per the US approved product label or in the opinion of the Investigator.
* Comorbid diagnosis of severe or very severe chronic obstructive pulmonary disease (COPD) per GOLD guidelines (GOLD 2021).
* Use of biologics that are approved for the treatment of asthma within 4 months or 5 half- lives (whichever is longer) prior to enrollment.
* Participation in an interventional clinical trial for asthma within 12 months prior to enrollment.
* Judgment by the Investigator that the participant is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Annualized asthma exacerbation rate (AAER) | Baseline period up to study Week 52
  Asthma exacerbation will be defined by worsening of asthma symptoms that leads to temporary bolus/burst of systemic corticosteroids for at least 3 consecutive days, or an emergency department (ED) or urgent care visit due to asthma that required systemic corticosteroid (SCS), and/or inpatient hospitalization (≥24 hours) due to asthma. The AAER is based on exacerbations reported by the investigator over 52 weeks.
  The exacerbation rate will be compared between the 12 month period before (baseline period) and the 12 month period after initiation of tezepelumab (up to study Week 52 - study period).
Proportion of participants with asthma exacerbations | Baseline period up to study Week 52
  The proportion of participants with asthma exacerbations in the 12 month periods before (baseline period) and after initiation of tezepelumab (study period) (up to study Week 52 - study period) will be assessed.
Proportion of participants who completed the 52 -week study period with any reduction in total number of asthma exacerbations | Baseline period up to study Week 52
  The proportion of participants who completed the 52 -week study period following tezepelumab initiation with any reduction, at least 50% reduction, and 100% reduction in total number of asthma exacerbations will be assessed.
Cumulative asthma exacerbation days | Baseline period up to study Week 52
  The cumulative asthma exacerbation days over 52 weeks before (baseline period) and after initiation of tezepelumab (study period) will be assessed.

SECONDARY OUTCOMES:
Time to first asthma exacerbation | Week 0 to Week 52
  The time to first exacerbation after initiation of tezepelumab will be assessed.
Rate of asthma exacerbations associated with hospitalizations | Baseline period up to study Week 52
  The rate of asthma exacerbations associated with hospitalization over 52 weeks before (baseline period) and after initiation of tezepelumab (study period) will be assessed.
Rate of asthma exacerbations associated with emergency department /urgent care (ED/UC) visits | Baseline period up to study Week 52
  The rate of asthma exacerbations associated with ED/UC visits over 52 weeks before (baseline period) and after initiation of tezepelumab (study period) will be assessed.
Rate of asthma exacerbations associated with hospitalizations or ED/UC visits over | Baseline period up to study Week 52
  The rate of asthma exacerbations associated with hospitalizations or ED/UC visits over 52 weeks before (baseline period) and after initiation of tezepelumab (study period) will be assessed.
Proportion of participants with asthma exacerbations associated with hospitalizations or ED/UC visits | Baseline period up to study Week 52
  The proportion of participants with asthma exacerbations associated with hospitalizations or ED/UC visits in in the 12-month periods before (baseline period) and after initiation of tezepelumab (study period) (up to study Week 52) will be assessed.
Cumulative asthma exacerbation days associated with hospitalizations or ED/UC visits | Baseline period up to study Week 52
  The cumulative asthma exacerbation days associated with hospitalizations or ED/UC over 52 weeks before (baseline period) and after initiation of tezepelumab (study period) will be assessed.
Pre-bronchodilator (pre-BD) forced expiratory volume in 1 second (FEV1) | Baseline (Week 0), Week 24, Week 52
  Lung function (FEV1) will be measured pre-bronchodilator (pre-BD) by spirometry test.
Change from baseline in pre-bronchodilator FEV1 | Baseline (Week 0), Week 24, Week 52
  Change from baseline in pre-bronchodilator FEV1 will be assessed as lung function parameters after initiation of tezepelumab.
Proportion of pre-BD FEV1 responders | Baseline (Week 0), Week 24, Week 52
  Proportion of pre-BD FEV1 responders is defined as participants who achieve either at least 5% or 100 mL improvement from baseline.
Asthma Control Questionnaire (ACQ-6) | Baseline (Week 0), Week 24, Week 52
  The ACQ-6 is a shortened version of the ACQ that assesses the adequacy of asthma control and change in asthma control which occurs spontaneously or as a result of treatment. ACQ assesses symptoms and rescue bronchodilator use.
  Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score is the mean of the responses.
Asthma Impairment and Risk Questionnaire (AIRQ) | Baseline (Week 0), Week 24, Week 52
  The Asthma Impairment and Risk Questionnaire (AIRQ) is a PRO tool intended to identify participants 12 years and older whose health may be at risk because of uncontrolled asthma.
  It has 10 questions that ask about respiratory symptoms, activity limitation, sleep, rescue medication use, social activities, exercise, difficulty controlling asthma, and exacerbations. All items have a yes/no response option and the tool is scored by summing the total number of 'yes' responses. This sum score is used to assess level of asthma control where: 0-1 is well controlled, 2-4 is not well controlled, and 5-10 is very poorly controlled. Thus, a higher score indicates worse control status.
St. George's Respiratory Questionnaire (SGRQ) | Baseline (Week 0), Week 24, Week 52
  The SGRQ is a 50-item PRO instrument developed to measure the health status of participants with airway obstruction diseases.
  The questionnaire is divided into 2 parts: part 1 consists of 8 items pertaining to the severity of respiratory symptoms in the preceding 4 weeks; part 2 consists of 42 items related to the daily activity and psychosocial impacts of the individual's respiratory condition. The SGRQ yields a total score and 3 components scores (symptoms, activity, and impacts). The total score indicates the impact of disease on overall health status. This total score is expressed as a percentage of overall impairment, in which 100 represents the worst possible health status and 0 indicates the best possible health status. Likewise, the domain scores range from 0 to 100, with higher scores indicative of greater impairment.
Change from baseline in ACQ-6 score | Baseline (Week 0), Week 24, Week 52
  Change from baseline in ACQ-6 score will be assessed.
Change from baseline in AIRQ score | Baseline (Week 0), Week 24, Week 52
  Change from baseline in AIRQ score will be assessed.
Change from baseline in SGRQ score | Baseline (Week 0), Week 24, Week 52
  Change from baseline in SGRQ score will be assessed.
Proportion of ACQ-6 responders | Baseline (Week 0), Week 24, Week 52
  ACQ-6 responders are defined as participants who achieve >=1 clinically important difference (MCID).
Proportion of AIRQ responders | Baseline (Week 0), Week 24, Week 52
  AIRQ responders is defined as participants who achieve ≥1 minimum clinically important difference (MCID).
Proportion of SGRQ responders | Baseline (Week 0), Week 24, Week 52
  SGRQ responders is defined as participants who achieve ≥1 minimum clinically important difference (MCID).
Proportion of participants who require any systemic corticosteroid (SCS) use | Baseline period up to study Week 52
  Proportion of participants who require any SCS use in the 12-month periods before (baseline period) and after initiation of tezepelumab (up to study Week 52 -study period) will be assessed.
Cumulative annualized SCS dose | Baseline period up to study Week 52
  Cumulative annualized SCS dose in the 12-month periods before (baseline period) and after initiation of tezepelumab (up to study Week 52- study period) will be assessed.
Proportion of participants who require longer-term (>30 consecutive days) SCS use | Baseline period up to study Week 52
  Proportion of participants who require longer-term (>30 consecutive days) SCS use in the 12-month periods before (baseline period) and after initiation of tezepelumab (up to study Week 52- study period) will be assessed.
Number and type of asthma-related healthcare resource utilization (HRU) | Baseline period up to study Week 52
  Number and type of asthma-related HRU in the 12-month period before (baseline period) and after initiation of tezepelumab (up to study Week 52- study period) will be assessed.
Duration of asthma-related hospitalizations | Baseline period up to study Week 52
  Duration of asthma-related hospitalization in the 12-month period before (baseline period) and after initiation of tezepelumab (up to study Week 52-study period) will be assessed.
AAER for asthma exacerbations (subgroups of participants) | Baseline period up to study Week 52
  The AAER based on asthma exacerbations in the 12-month period before (baseline period) and after initiation of tezepelumab (up to study Week 52- study period) will be assessed in the following subgroups of participants: Blood eosinophil count (BEC) ≥300 cells/microliter; BEC <300 cells/microliter; With a clinically-relevant allergy to a perennial aeroallergen; Without a clinically-relevant allergy to a perennial aeroallergen; Participants who identify as Black/African American; Adolescents (12-17 years); Comorbid diagnosis of mild to moderate COPD; Significant smoking history (≥10 pack-years of smoking).
Proportion of participants with asthma exacerbations (subgroups of participants) | Baseline period up to study Week 52
  The proportion of participants with asthma exacerbations in the 12-month period before (baseline period) and after initiation of tezepelumab (up to study Week 52- study period) will be assessed in the following subgroups of participants: BEC ≥300 cells/microliter; BEC <300 cells/microliter; With a clinically-relevant allergy to a perennial aeroallergen; Without a clinically-relevant allergy to a perennial aeroallergen; Participants who identify as Black/African American; Adolescents (12-17 years); Comorbid diagnosis of mild to moderate COPD; Significant smoking history (≥10 pack-years of smoking).
Proportion of participants who completed the 52 -week study with any reduction in total number of asthma exacerbations (subgroups of participants) | Week 0 to Week 52
  The proportion of participants who completed the 52 -week study period following tezepelumab initiation with any reduction, at least 50% reduction, and 100% reduction in total number of asthma exacerbations will be assessed in the following subgroups of participants: BEC ≥300 cells/microliter; BEC <300 cells/microliter; With a clinically-relevant allergy to a perennial aeroallergen; Without a clinically-relevant allergy to a perennial aeroallergen; Participants who identify as Black/African American; Adolescents (12-17 years); Comorbid diagnosis of mild to moderate COPD; Significant smoking history (≥10 pack-years of smoking).
Cumulative asthma exacerbation days (subgroups of participants) | Baseline period up to study Week 52
  The cumulative asthma exacerbation days over 52 weeks before (baseline period) and after initiation of tezepelumab (study period) will be assessed in the following subgroups of participants: BEC ≥300 cells/microliter; BEC <300 cells/microliter; With a clinically-relevant allergy to a perennial aeroallergen; Without a clinically-relevant allergy to a perennial aeroallergen; Participants who identify as Black/African American; Adolescents (12-17 years); Comorbid diagnosis of mild to moderate COPD; Significant smoking history (≥10 pack-years of smoking).
Rate of asthma exacerbations associated with hospitalizations (subgroups of participants) | Baseline period up to study Week 52
  The rate of asthma exacerbations associated with hospitalization over 52 weeks before (baseline period) and after initiation of tezepelumab (study period) will be assessed in the following subgroups of participants: BEC ≥300 cells/microliter; BEC <300 cells/microliter; With a clinically-relevant allergy to a perennial aeroallergen; Without a clinically-relevant allergy to a perennial aeroallergen; Participants who identify as Black/African American; Adolescents (12-17 years); Comorbid diagnosis of mild to moderate COPD; Significant smoking history (≥10 pack-years of smoking).
Rate of asthma exacerbations associated with emergency department urgent care (ED/UC) visits (subgroups of participants) | Baseline period up to study Week 52
  The rate of asthma exacerbations associated with ED/UC visits over 52 weeks before (baseline period) and after initiation of tezepelumab (study period) will be assessed in the following subgroups of participants: BEC ≥300 cells/microliter; BEC <300 cells/microliter; With a clinically-relevant allergy to a perennial aeroallergen; Without a clinically-relevant allergy to a perennial aeroallergen; Participants who identify as Black/African American; Adolescents (12-17 years); Comorbid diagnosis of mild to moderate COPD; Significant smoking history (≥10 pack-years of smoking).
Rate of asthma exacerbations associated with hospitalizations or ED/UC visits over (subgroups of participants) | Baseline period up to study Week 52
  The rate of asthma exacerbations associated with hospitalizations or ED/UC visits over 52 weeks before (baseline period) and after initiation of tezepelumab (study period) will be assessed in the following subgroups of participants: BEC ≥300 cells/microliter; BEC <300 cells/microliter; With a clinically-relevant allergy to a perennial aeroallergen; Without a clinically-relevant allergy to a perennial aeroallergen; Participants who identify as Black/African American; Adolescents (12-17 years); Comorbid diagnosis of mild to moderate COPD; Significant smoking history (≥10 pack-years of smoking).
Number and type of asthma-related HRU (subgroups of participants) | Baseline period up to study Week 52
  Number and type of asthma related HRU in the 12-month period before (baseline period) and after initiation of tezepelumab (up to study Week 52- study period) will be assessed in the following subgroups of participants: BEC ≥300 cells/microliter; BEC <300 cells/microliter; With a clinically-relevant allergy to a perennial aeroallergen; Without a clinically-relevant allergy to a perennial aeroallergen; Participants who identify as Black/African American; Adolescents (12-17 years); Comorbid diagnosis of mild to moderate COPD; Significant smoking history (≥10 pack-years of smoking).
Duration of asthma-related hospitalizations (subgroups of participants) | Baseline period up to study Week 52
  Duration of asthma-related hospitalization in the 12- month period before (baseline period) and after initiation of tezepelumab (up to study Week 52- study period) will be assessed in the following subgroups of participants: BEC ≥300 cells/microliter; BEC <300 cells/microliter; With a clinically-relevant allergy to a perennial aeroallergen; Without a clinically-relevant allergy to a perennial aeroallergen; Participants who identify as Black/African American; Adolescents (12-17 years); Comorbid diagnosis of mild to moderate COPD; Significant smoking history (≥10 pack-years of smoking).

OTHER OUTCOMES:
Number of participants with serious adverse events, adverse events that lead to tezepelumab treatment discontinuation, and adverse events of special interest | Week 0 to Week 52
  The safety and tolerability of tezepelumab will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Njira Lugogo., MD., Principal Investigator — University of Michigan Health. Michigan, USA
Locations (37):
- United States (37):
  - Research Site, Mobile, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Rancho Mirage, California
  - Research Site, Westminster, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Chicago, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Upper Marlboro, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Saint Paul, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Hollis, New York
  - Research Site, Horseheads, New York
  - Research Site, Rochester, New York
  - Research Site, Valhalla, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Altoona, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Greenville, South Carolina
  - Research Site, Hendersonville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Lugogo NL, Akuthota P, Sumino K, Mathur SK, Burnette AF, Lindsley AW, Llanos JP, Marchese C, Ambrose CS, Emmanuel B. Effectiveness and Safety of Tezepelumab in a Diverse Population of US Patients with Severe Asthma: Initial Results of the PASSAGE Study. Adv Ther. 2025 Jul;42(7):3334-3353. doi: 10.1007/s12325-025-03231-6. Epub 2025 May 19. PMID 40388086